CLINICAL TRIAL: NCT05914896
Title: Hyperosmolar Priming Solution for Cardiopulmonary Bypass May Increase the Risk for Postoperative Acute Kidney Injury: Results From Double-blinded Randomised Controlled Trial
Brief Title: Hyperosmolality and Acute Kidney Injury After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UmeaU-OSM
Record Dates: First submitted 2023-06-07; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Acute Kidney Injury; Osmolality Disturbance; Cardiopulmonary Bypass
Keywords: Cardiopulmonary Bypass; Priming Solution; Plasma Osmolality; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Randomisation into two groups based on the osmolality level in the priming solution used for cardiopulmonary bypass.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Priming of the heart-lung machine performed by a staff member not affiliated to the study protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NormOsmo (No Intervention): This group received a priming solution with normal osmolality.
- HighOsmo (Active Comparator): This group received a priming solution with high osmolality
  Interventions: Drug: HighOsmo

INTERVENTIONS:
Drug: HighOsmo — This group received a priming solution with high osmolality
  Arms: HighOsmo

SUMMARY:
The goal of this randomized controlled trial is to test if a hyperosmolar prime solution used for cardiopulmonary bypass increases the risk for acute postoperative kidney injury.

DETAILED DESCRIPTION:
Two-hundred cardiac surgical patients were randomised into two groups based on the osmolality level of the prime solution used for cardiopulmonary bypass. The high osmolality group (966 mOsm) received a prime solution containing Ringer-Acetate 1000 ml + Mannitol 400 ml (60 g) + Sodium-Chloride 40 ml (160 mmol) and Heparin 2 ml (10 000 IU), while the reference group with normal osmolality (388 mOsm) received a prime solution containing Ringer-Acetate 1400 ml and Heparin 2 ml (10 000 IU).

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for routine cardiac surgical procedures requiring cardiopulmonary bypass.

Exclusion Criteria:

* Patients requiring acute surgical intervention within 24 h or profound hypothermia during surgery were excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Postoperative Acute Kidney Injury | Three days
  Defined according to the KDIGO definition

CONTACTS AND LOCATIONS:
Overall Officials: Staffan Svenmarker, PhD, Principal Investigator — Public Health & Clinical Medicine Umeå University, Sweden
Locations (1):
- Department of Public Health Clinical Medicine Umeå University, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No
Limited by ethical regulations

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152